CLINICAL TRIAL: NCT02445872
Title: Safety and Efficacy of Aprepitant for Chemotherapy-Induced Nausea and Vomiting in Patients With Lung Cancer Receiving Multiple-day Cisplatin Chemotherapy
Brief Title: Safety and Efficacy of Aprepitant for CINV in Patients With Lung Cancer Receiving Multiple-day Cisplatin Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Qiong Zhao, Chief, Department of Thoracic Oncology, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZYTOP1502
Record Dates: First submitted 2015-04-05; First posted 2015-05-15 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting; Lung Cancer
Keywords: Nausea; Vomiting; Chemotherapy-induced Nausea and Vomiting; CINV; Aprepitant; Lung cancer
MeSH Terms: conditions — Vomiting; Lung Neoplasms; Nausea | interventions — Aprepitant; Palonosetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Aprepitant: 125mg PO on day1, 80mg PO on day2 and day3. Palonosetron (a 5-HT3 receptor antagonist): 0.25 mg IV push on day 1 only. Dexamethasone: 5mg IV push once daily from day 1 to day 3,and 3.75mg PO on days 4-5.
  Interventions: Drug: Aprepitant; Drug: Palonosetron; Drug: Dexamethasone
- Arm B (Active Comparator): Palonosetron: 0.25 mg IV push on day 1 only. Dexamethasone: 5mg IV push once daily from day 1 to day 3,and 7.5mg PO on days 4-5.
  Interventions: Drug: Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Aprepitant — Aprepitant:The first day, one 125 mg capsule will be administered per oral, 1 hour before chemotherapy. Thereafter one 80 mg capsule will be repeated daily between 8 to 10 a.m. during days 2 to 3
  Other Names: Emend
  Arms: Arm A
Drug: Palonosetron
Drug: Dexamethasone

SUMMARY:
Aprepitant is an oral neurokinin-1(NK-1) antagonist which is used for the prevention of chemotherapy-induced nausea and vomiting (CINV). This phase II clinical trial was designed to evaluate the efficacy of aprepitant in the prevention of CINV with lung cancer patients receiving 3-day cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
Patients pathologic diagnosed of advanced non-small cell lung cancer, according to NCCN non-small cell lung cancer guide line(2015 V1).The patient should receive a 3-day cisplatin-based chemotherapy, are randomized divided into two groups, aprepitant group and placebo group. In aprepitant group, patients would receive aprepitant(125 mg po at day1, 80 mg at day2-3) combination with palonosetron and dexamethasone(5mg iv at day1-3, 3.75mg po at day4-5). In placebo group patients would receive palonosetron and dexamethasone(5mg iv at day1-3, 7.5mg po at day4-5).During the treatment, any grade of nausea and vomiting should be recorded in order to evaluate the complete response rate of CINV, other side-effects should be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who was confirmed lung cancer by pathologic histology or cytology.
2. Males or females aged ≥18 years, <80 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Life expectancy ≥12 weeks.
4. Males and females should be contraceptive during the period of the trial until 8 weeks after the last administration of the drug.
5. Patients with asymptomatic, treated brain metastases are eligible for trial participation.
6. Adequate bone marrow, renal, and liver function are required.
7. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
8. Institutional review board-approved informed consent will be obtained for every patient before initiation of any trial-specific procedure or treatment.

Exclusion Criteria:

1. History of sensitivity/idiosyncrasy to aprepitant or excipients
2. Condition that might interfere with drug absorption, distribution metabolism or excretion.
3. Concomitant use of agents that are known to interfere with aprepitant pharmacokinetics
4. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
5. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
6. Female subjects should not be pregnant or breast-feeding.
7. Inadequate hematological function.
8. Abnormal liver and renal function.
9. Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 5 days after the end of chemotherapy
  The primary endpoint is the overall rate of patients achieving a complete response (defined as no emetic episode and no use of rescue medication) during the overall phase

SECONDARY OUTCOMES:
Complete Control (No emetic episode, no need for rescue medication, with a maximum grade of mild nausea) | 5 days after the end of chemotherapy
  No emetic episode, no need for rescue medication, with a maximum grade of mild nausea
Emesis-free | 5 days after the end of chemotherapy
  Percentage of patients without emetic episodes
Presence of nausea | 5 days after the end of chemotherapy
  Presence of nausea graded according to Likert scale (none, mild, moderate and severe)
Safety and tolerability (adverse events related to study drug administration) | 5 days after the end of chemotherapy
  Number of patients experienced at least one adverse events related to study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Gao HF, Liang Y, Zhou NN, Zhang DS, Wu HY. Aprepitant plus palonosetron and dexamethasone for prevention of chemotherapy-induced nausea and vomiting in patients receiving multiple-day cisplatin chemotherapy. Intern Med J. 2013 Jan;43(1):73-6. doi: 10.1111/j.1445-5994.2011.02637.x. PMID 22141732